CLINICAL TRIAL: NCT07145450
Title: Phase 1/2 Master Protocol for Open-Label, Multi-Centre, Single-Arm Sub-Studies, First in Human Clinical Studies of TCR-T Therapy (Autologous TCR- Modified T-Cell Therapy) Targeting Mutated Kirsten Rat Sarcoma (mutKRAS) Administered in Metastatic or Locally Advanced Pancreatic Ductal Adenocarcinoma (PDAC) Adult Patients With Specific mutKRAS and Human Leukocyte Antigen (HLA) Genotypes
Brief Title: Master Protocol of TCR-modified T Cell Therapy Targeting HLA-restricted KRAS Antigen Administered in Adult Patients With Metastatic or Locally Advanced PDAC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anocca AB (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP-ANOC-IS-001
Record Dates: First submitted 2025-07-09; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: PDAC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ANOC-001 (Other): Treatment
  Interventions: Biological: ANOC-001 (TCR-T cells targeting KRAS G12V mutation presented by specific HLA alleles)
- ANOC-002 (Other): Treatment
  Interventions: Biological: ANOC-002 (TCR-T cells targeting KRAS G12V mutation presented by specific HLA alleles)
- ANOC-003 (Other): Treatment
  Interventions: Biological: ANOC-003 (TCR-T cells targeting KRAS G12D mutation presented by specific HLA alleles)

INTERVENTIONS:
Biological: ANOC-001 (TCR-T cells targeting KRAS G12V mutation presented by specific HLA alleles) — The cells will be gene edited and administered by a single IV infusion on Day 1.
  Drugs: Cyclophosphamide and Fludarabine will be used as a lymphodepleting chemotherapy.
  Arms: ANOC-001
Biological: ANOC-002 (TCR-T cells targeting KRAS G12V mutation presented by specific HLA alleles) — The cells will be gene edited and administered by a single IV infusion on Day 1. Drugs: Cyclophosphamide and Fludarabine will be used as a lymphodepleting chemotherapy.
  Arms: ANOC-002
Biological: ANOC-003 (TCR-T cells targeting KRAS G12D mutation presented by specific HLA alleles) — The cells will be gene edited and administered by a single IV infusion on Day 1. Drugs: Cyclophosphamide and Fludarabine will be used as a lymphodepleting chemotherapy
  Arms: ANOC-003

SUMMARY:
This is an open-label, multi-centre, single-arm Phase 1/2 clinical trial of the safety, expansion, persistence and clinical activity of a set of engineered autologous T cells products each capable of recognizing a specific combination mutated KRAS and HLA, activating the T cells and exerting anti- tumour activity in patients with metastatic or locally advanced PDAC.

DETAILED DESCRIPTION:
This is a phase 1/2 study of engineered autologous T cells (TCR targeting KRAS G12V (ANOC-001 sub-study 1), (ANOC-002 sub-study 2) and KRAS 12D (ANOC-003 sub-study 3) capable of recognizing the tumour antigen(s), activating the T cells and exerting anti-tumour activity in patients with metastatic or locally advanced PDAC following a SoC first-line therapy.

The protocol procedures will be performed in two parts. Part 1 includes pre- screening/screening eligibility, enrolment and leukapheresis. Part 2 includes lymphodepletion, TCR-T cell infusion and all study assessments until the end-of-treatment or early discontinuation .

In the dose escalation part of each sub-study, two doses will be assessed in a classical 3+3 dose escalation design to assess the safety and tolerability of TCR-T cells with the goal to identify the optimal safe dose for each product.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (18 years or older) with newly diagnosed metastatic PDAC or locally advance PDAC disease.
2. HLA genotyping confirmed with a high-resolution method.
3. Confirmed KRAS G12V or KRAS G12D mutation in tumour using biopsy sample.
4. Fertile male and female patients must use a highly effective contraceptive method before, during, and for at least 6 months after the last mutKRAS TCR infusion. Acceptable contraception for women includes implants, injectables, combined oral contraceptives, intrauterine devices (IUDs), sexual abstinence, or a partner who has been vasectomized for at least 6 months. Acceptable contraception for male includes having had a vasectomy for at least 6 months, sexual abstinence, to condoms plus spermicide. Fertile female and male patients must adhere to any treatment-specific pregnancy prevention guidelines for cyclophosphamide (refer to SmPC).
5. Confirmed clinical benefit to SoC treatments and absence of disease progression according to the PI judgement.
6. Measurable disease by RECIST 1.1 criteria at the time of first treatment. Baseline imaging (for example, diagnostic CT chest/abdomen/pelvis and imaging of the affected extremity or brain, as appropriate), magnetic resonance imaging (MRI or CT scan) must be obtained within 8 weeks of the first planned T cell infusion. CT can be substituted for MRI in patients unable to have CT contrast.

Exclusion Criteria:

1. Another malignancy other than PDAC.
2. Current or history of brain metastasis.
3. Patient with known genetic status for whom other treatments are available e.g. BRCA, MSI-H.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2030-04-02 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1-Proportion of participants with dose limiting toxicity of ANOC-001, ANOC-002 and ANOC-003, graded according to American Society of Transplantation and Cellular Therapy (ASTCT) consensus criteria. | First infusion through Day 28
Phase 1-Number of participants with adverse events graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), v5.0. | First infusion through Day 28
Phase 1- Identification of the Maximum tolerated dose/Maximum administered dose and Recommended Phase 2 Dose of ANOC-001/ANOC-002/ANOC-003 cells that can be administered safely in patients with metastatic and locally advanced PDAC. | First infusion through Day 28
Phase 2-Number of participants with adverse events of special interest (AESI) according to NCI CTCAE v5.0. | Baseline through 24 months post-treatment
Phase 2- Proportion of participants with Objective Response Rate (ORR) defined as the number of patients with a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) per RECIST v1.1 divided by the number of treated patients. | Baseline through 24 months post-treatment
Phase 2-Proportion of participants with Clinical benefit rate (CBR) defined as percentage of patients with stable disease (SD) more than 3 months, or PR/CR from the time of study treatment. | Baseline through 24 months post-treatment
Phase 2-Proportion of participants with Clinical benefit determined by the investigator, assessed anytime at 8- to 12-week intervals post TCR-T cell infusion. | Baseline through 24 months post-treatment

SECONDARY OUTCOMES:
Phase 1 and Phase 2: Percentage of patients who receive protocol-defined target dose of ANOC-001, ANOC-002 and ANOC-003. | From leukapheresis through product release and infusion (Day 1), on an average of 2-4 months for each participant
Phase 1 and Phase 2: Proportion of investigational product- ANOC-001, ANOC-002 and ANOC-003 that comply with the specifications as compared to the total number of the IMP manufactured | From leukapheresis through product release and infusion (Day 1), on an average of 2-4 months for each participant
Phase 1 and Phase 2-Maximum expansion and persistence of TCR T cells following infusion by quantitative PCR | Baseline through 24 months post-treatment
Phase 1 and Phase 2- Proportion of participants achieving Progression Free Survival (PFS) defined as the time from study treatment to the first occurrence of disease progression or death, whichever occurs first. | Baseline through 24 months post-treatment
Phase 1 and Phase 2- Proportion of participants achieving Overall Survival (OS) defined as the time from study treatment to death from any cause. | Baseline through 24 months post-treatment
Phase 1 and Phase 2- Proportion of participants achieving Duration of Response (DoR) defined as the time from study treatment to disease progression or death in patients who achieve CR or PR. | Baseline through 24 months post-treatment

OTHER OUTCOMES:
Exploratory-Phase 1 and 2-To evaluate correlation of T cell persistence with safety and clinical response and with phenotype of infused T cells | Baseline through 24 months post-treatment
Exploratory-Phase 1 and 2-To evaluate types and levels of cytokines in peripheral blood | Baseline through 24 months post-treatment
Exploratory-Phase 1 and 2-To evaluate change in ctDNA and CTC/exosome load | Baseline through 24 months post-treatment
Exploratory-Phase 1 and 2-Conventional serum markers e.g., CA19-9, CEA will be tested locally | Baseline through 24 months post-treatment
Exploratory-Phase 1 and 2-CD8 ImmunoPET imaging will be considered as an ad-hoc basis to assess TCR-T cell immune infiltration into primary tumour and metastases | Baseline through 24 months post-treatment
Exploratory-Phase 1 and 2-To evaluate longitudinal biopsy if possible to study the TME by the means of immunohistochemistry (IHC) and RNA-bulk sequencing methods. | Baseline through 24 months post-treatment

CONTACTS AND LOCATIONS:
Locations (8):
- Herlev and Gentofte University Hospital, Copenhagen, Denmark
- Germany (4):
  - Charité Universitätsmedizin Berlin, Berlin
  - Technische Universitaet Dresden - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinikum Heidelberg, Heidelberg
  - University Hospital and Faculty of Medicine Eberhard Karls University Tübingen, Tübingen
- Netherlands (2):
  - Amsterdam UMC - VU Medical Center, Amsterdam
  - Radboud University Medical Center, Nijmegen
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No